CLINICAL TRIAL: NCT02162576
Title: Asthma Data Innovation Demonstration Project: Impact of a Mobile Health, Sensor-driven Asthma Management Platform on Asthma Symptoms, Control and Self-management
Brief Title: Asthma Data Innovation Demonstration Project
Acronym: ADID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Van Sickle (Industry)
Collaborators: Foundation for a Healthy Kentucky (Other); Norton Healthcare Foundation (Other); Owsley Brown Charitable Foundation (Unknown)
Responsible Party: Sponsor-Investigator, David Van Sickle, CEO, Reciprocal Labs
Organization: Reciprocal Labs (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH LVL - 40202
Record Dates: First submitted 2014-06-06; First posted 2014-06-12 (Estimated); Results first posted 2017-12-26 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases; Respiratory Hypersensitivity; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases
Keywords: asthma; asthma control; healthcare utilization costs; community hotspots; public health research
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases; Respiratory Hypersensitivity; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Propeller Health intervention group (Other): All participants attached the Propeller sensor to their SABA medications and tracked the time and location of use for up to 13 months, to capture seasonal variation in medication use, symptoms and environmental triggers. The first 30-day run-in period served as a control period to assess levels of asthma control and SABA use; subject actuations were tracked, but participants and physicians did not receive their data or feedback. After the run-in period, participants received the full intervention for 12 months (see intervention for description).
  Interventions: Device: Propeller Health intervention

INTERVENTIONS:
Device: Propeller Health intervention — The Propeller intervention works through the provision of information to patients and their providers. With the Propeller sensor device in place, each actuation of a patient's rescue inhaler is recorded with an automatic time stamp and geographic location. Actuation data are then securely transmitted to Propeller Health where the information is also compiled into individual reports via mobile apps, online dashboards, email reports and text message reminders that are returned to the patient. This communication provides an ongoing assessment of their management based on the national guidelines, together with personalized information to help encourage and support self-management. Each participant was invited to share reports with his or her healthcare provider, but this was not required.
  Other Names: Asthmapolis

SUMMARY:
Propeller Health is collaborating with the City of Louisville and other local partners to carry out a focused demonstration project that will evaluate the effectiveness of the Propeller Health approach to asthma management while exploring means to use real-time data on asthma exacerbations in a public health setting. The Asthma Data Innovation Demonstration Project (ADID) will use wireless sensor technology to develop spatial and temporal data on the use of rescue inhalers by 120 study subjects with asthma in the Louisville metropolitan area. Propeller Health will process these data to support two general strategies.

Asthma self management: Rescue inhaler actuation data will be compiled into individualized feedback reports to support asthma self management. Propeller Health will combine information on individual rescue inhaler actuations with evidence-based asthma management tips into real-time reports that will be provided to subjects. ADID staff will evaluate any resulting improvements in asthma control that may be based on this information. Subjects may share reports with their healthcare providers.

Municipal purposes: The second strategy is to provide aggregated and de-identified, spatial and temporal asthma rescue inhaler actuation data to City personnel and authorized public health researchers in Louisville. These data will show the times and locations of the use of rescue inhalers by the 120 study subjects throughout the greater Louisville area. ADID staff will work with City personnel and researchers to investigate how this unprecedented level of detailed information on exacerbations can be used best to increase public awareness of environmental triggers while supporting public health surveillance efforts around respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported provider diagnosis of asthma
* Prescription for Short Acting Beta Agonist (SABA) at study intake

Exclusion Criteria:

* Subject is under the age of 5 at the beginning of the study
* Subject does not speak English
* Subject does not have access to the Internet or email to receive reports
* Subject has substantial co-morbidity (self-reported provider diagnosis of COPD)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2012-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Van Sickle, PhD, Principal Investigator — Propeller Health
Locations (1):
- Jefferson County, Louisville, Kentucky, United States

REFERENCES:
- [Result] Barrett M, Combs V, Su JG, Henderson K, Tuffli M; AIR Louisville Collaborative; AIR Louisville Collaborative. AIR Louisville: Addressing Asthma With Technology, Crowdsourcing, Cross-Sector Collaboration, And Policy. Health Aff (Millwood). 2018 Apr;37(4):525-534. doi: 10.1377/hlthaff.2017.1315. PMID 29608361
- [Result] Barrett MA, Humblet O, Marcus JE, Henderson K, Smith T, Eid N, Sublett JW, Renda A, Nesbitt L, Van Sickle D, Stempel D, Sublett JL. Effect of a mobile health, sensor-driven asthma management platform on asthma control. Ann Allergy Asthma Immunol. 2017 Nov;119(5):415-421.e1. doi: 10.1016/j.anai.2017.08.002. PMID 29150069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited residents from community events, clinics and retail pharmacies using a convenience sampling strategy. Participants were eligible if they reported a physician diagnosis of asthma and a current prescription for SABA medication. Recruitment occurred between 6/2012 and 1/2013, with the last subject exiting the program in 1/2014.
Pre-assignment Details: A run-in period of 30 days was designed to limit enrollment to those participants who could comply with the study requirements. In order to be included in the study, the participant would have to 1) create an account, 2) activate their sensor, and 3) remain active (defined by sensor syncing) for the first 30 day run-in period.
Groups:
- Propeller Health Intervention Group: All participants attached the Propeller sensor to their SABA medications and tracked the time and location of use for up to 13 months, to capture seasonal variation in medication use, symptoms and environmental triggers. The first 30-day run-in period served as a control period to assess levels of asthma control and SABA use; subject actuations were tracked, but participants and physicians did not receive their data or feedback. After the run-in period, participants received the full intervention for 12 months.
  The Propeller sensor passively records inhaler actuations with a time stamp and location. Actuation data are then securely transmitted to Propeller Health where the information is also compiled into individual reports via multiple platforms, providing an assessment of their management based on the national guidelines, together with personalized information to help encourage and support self-management (see intervention description for full details).
Period: Overall Study
Arm/Group | Propeller Health Intervention Group
Started | 95
Completed | 95
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 95 participants were enrolled in the study program.
Arm/Group | Propeller Health Intervention Group
Number analyzed (Participants) | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42
  Between 18 and 65 years | 51
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (18.3)
Sex/Gender, Customized [Number; unit: participants]
  Female | 53
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 95
Asthma Control Test [Mean (Standard Deviation); unit: units on a scale] — ACT is a patient self-administred tool for identifying those with poorly controlled asthma. There are 5 items, with 4-week recall, that address symptoms and daily functioning topics. Each item is measured on 5-point scale. The ACT score ranges from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
  units on a scale | 17.51 (4.45)

OUTCOME MEASURES:

1. Primary Outcome: Change in Rescue Inhaler Actuations/Person/Day
Description: The Propeller Health sensor permits the capture of objective time and location data on each actuation of the rescue inhaler. The mean number of rescue inhaler events per participant per day will be assessed for each day in the study, and the difference between the baseline month and all subsequent months will be evaluated.
Time Frame: Change from baseline to study exit, up to 13 months
Measure: Mean (Standard Deviation); unit: puffs per participant per day
Arm/Group | Propeller Health Intervention Group
Number analyzed (Participants) | 95
puffs per participant per day | -0.37 (0.27)

2. Secondary Outcome: Percent Change in the Proportion of Participants With an Asthma-free Day
Description: Each 24-hour period without an actuation of a rescue inhaler was counted as an asthma-free day. The proportion of participants with an asthma-free day was calculated for each day of the program, with the denominator including all active participants on that day of the program, defined as those that synced after that date.
Time Frame: Change from baseline period to study exit (approximately 13 months)
Measure: Number; unit: percentage change
Groups:
- Propeller Health Intervention: All participants attached the Propeller sensor to their SABA medications and tracked the time and location of use for up to 13 months, to capture seasonal variation in medication use, symptoms and environmental triggers. The first 30-day run-in period served as a control period to assess levels of asthma control and SABA use; subject actuations were tracked, but participants and physicians did not receive their data or feedback. After the run-in period, participants received the full intervention for 12 months.
  The Propeller sensor passively records inhaler actuations with a time stamp and location. Actuation data are then securely transmitted to Propeller Health where the information is also compiled into individual reports via multiple platforms, providing an assessment of their management based on the national guidelines, together with personalized information to help encourage and support self-management (see intervention description for full details).
Arm/Group | Propeller Health Intervention
Number analyzed (Participants) | 95
percentage change | 23

3. Secondary Outcome: Percent Change in the Proportion of Participants With Well-controlled Asthma
Description: Daily control status was assessed based upon the timing and frequency of SABA actuations according to NAEPP guidelines. The proportion of the study cohort defined as well controlled, not well controlled and poorly controlled was assessed weekly throughout the program.
Time Frame: Baseline and study exit (approximately 13 months)
Measure: Number; unit: percent change
Arm/Group | Propeller Health Intervention
Number analyzed (Participants) | 95
percent change | 33

ADVERSE EVENTS:
Groups:
- Propeller Health Intervention: After the control period is completed at 1 month, all participants will continue using their sensors, and will begin to receive the full intervention for 12 months. The intervention includes access to all of the participant's sensor-collected data, trends, educational information and weekly reports. The 13-month term was chosen in order to eliminate any seasonal variation in asthma exacerbations.
  Propeller Health: The digital sensor records rescue inhaler actuations, as well as time and date stamp, and location if available. Actuation data are then securely transmitted to Propeller Health where events and an assessment of asthma control can be viewed in secure online interfaces. The information is also compiled into individual reports via mobile apps, online dashboards, email reports and text message reminders that are returned to the patient. Each participant was invited to share reports with his or her healthcare provider, but this was not required.
Arm/Group | Propeller Health Intervention
Serious Adverse Events (participants affected / at risk) | 0/95
Other Adverse Events (participants affected / at risk) | 0/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No